CLINICAL TRIAL: NCT06203704
Title: OPTIMISE-CKD CEE: A Multinational, Observational, Secondary Data Study Describing Management and Treatment With Dapagliflozin in Routine Clinical Practice Among Patients With Chronic Kidney Disease in Central Eastern Europe
Brief Title: Observational Secondary Data Study Describing Treatment With Dapagliflozin Among Adult Chronic Kidney Disease Patients
Acronym: OPTIMISE-CKD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D169AR00025
Record Dates: First submitted 2023-12-12; First posted 2024-01-12 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
The OPTIMISE-CKD CEE study design will create a real-world evidence platform that systematically leverages the routine data collection made by Investigators and will help obtain relevant insights from clinical practice. This study is likely to include a more heterogeneous population compared with the constraints required by interventional study protocols. Treatment decisions, clinical outcomes, and common treatment scenarios in the context of routine care of CKD are likely to be more generalizable than those from clinical trials.

It is important to assess the current CKD treatment with dapagliflozin. The research questions can be divided into two categories:

1. What does the dapagliflozin utilisation in CKD look like?

   a. Who are being treated?
2. What are the selected outcomes of interest and treatment patterns among CKD patients treated with dapagliflozin, with or without type 2 diabetes (T2D) up to 12 months post-initiation?

Primary objective is to characterize dapagliflozin utilisation in clinical practice, by describing treatment naïve patients who are treated with dapagliflozin for CKD.

Secondary objectives are to describe selected outcomes of interest and treatment patterns among CKD patients treated with dapagliflozin up to 12 months post-initiation.

The OPTIMISE-CKD CEE study is a multinational, observational, longitudinal cohort study, with a pre-post design, which will include patients who are treated with dapagliflozin with CKD in real-world clinical practice, utilising secondary data sources. This is a secondary data collection study, where variables are extracted from electronic or paper medical records.

Seven Central Eastern Europe countries are planned to participate in the study: Bulgaria, Croatia, Hungary, Poland, Romania, Serbia and Slovenia. A total number of 1090 patients are estimated to be included in the study.

The study population will consist of adult patients with CKD who meet the country-specific label for dapagliflozin as treatment for CKD across CEE.

DETAILED DESCRIPTION:
The OPTIMISE-CKD CEE study design will create a real-world evidence platform that systematically leverages the routine data collection made by Investigators and will help obtain relevant insights from clinical practice. This study is likely to include a more heterogeneous population compared with the constraints required by interventional study protocols. Treatment decisions, clinical outcomes, and common treatment scenarios in the context of routine care of CKD are likely to be more generalizable than those from clinical trials. The results of the study will be used to better inform the medical community, and decision-makers about current and future needs in the CKD management in CEE in real-life setting. The approved label encompasses all CKD patients at risk of disease progression and is thereby broader than the DAPA-CKD trial population. It is important for physicians and patients to better understand dapagliflozin use in CKD in routine clinical practice, particularly among patients who might have been underrepresented in clinical trials. Additionally, payers require additional evidence from the broader CKD population prior to making reimbursement recommendations that will enable access for all patients who have the approved CKD indication.

It is important to assess the current CKD treatment with dapagliflozin. Primary objective is to characterize dapagliflozin utilisation in clinical practice, by describing treatment naïve patients who are treated with dapagliflozin for CKD.

To describe characteristics among patients newly initiated on dapagliflozin 10 mg for CKD, the following will be used:

1. Baseline demographics and clinical characteristics
2. Baseline laboratory measures
3. Baseline concomitant medications, by drug class and specific drugs of interest.

Secondary objectives are to describe selected outcomes of interest and treatment patterns among CKD patients treated with dapagliflozin up to 12 months post-initiation:

1. CKD progression (advancement in CKD stage)
2. Selected clinical outcomes: cardio-renal events (e.g., CKD progression, HF, nonfatal stroke, nonfatal MI)
3. Selected healthcare resource utilization, e.g., all-cause hospitalizations, cardio-renal hospitalizations (CKD, hHF, MACE [nonfatal stroke, nonfatal MI])
4. Treatment patterns of dapagliflozin, RAASi (ACE inhibitors / ARB), and other selected medications used for CVD and T2D, defined as time to discontinuation (dapagliflozin only), medication additions, discontinuations, and dosage changes.

Study design: The OPTMISE-CKD CEE regional study is an observational, longitudinal cohort study with a pre-post design, which will include patients who are treated with dapagliflozin for CKD in real-world clinical practice, utilising secondary data sources in 7 countries (Bulgaria, Croatia, Hungary, Poland, Romania, Serbia and Slovenia) from CEE. The data extraction from medical charts will be made by Investigators, only after eligible patients express their written consent for data collection in the OPTIMISE-CKD study during the enrolment period defined at study level. A period of min. 30 days and max. 90 days after dapagliflozin was initiated is required for enrolment. Given the secondary data collection character of this study, no study-specific diagnostic and monitoring processes are to be applied to the patients.

Data Sources: Disease and treatment-related information routinely collected in clinical practice will be extracted by Investigators from paper and/or electronic health records (EHR). Data from all participating centers will be collected into a single anonymized dataset for analysis, by means of electronic case report forms (CRFs).

Study Population: Adult patients (aged ≥18 years) with CKD who initiated dapagliflozin 10 mg and meet all inclusion criteria and none of the exclusion criteria. Enrolment is to be performed minimum 30 days and maximum 90 days since initiation of dapagliflozin for CKD. Previous treatment with dapagliflozin or SGLT-2i deems patient ineligibility.

Exposure(s): The study will describe CKD treatments and drug utilisation patterns (Section 4.2), specifically for dapagliflozin 10 mg, RAASi and other treatments routinely used in the management of CKD patients (see Section 4.4) up to 12 months post-dapagliflozin initiation. Data on exposure to dapagliflozin, RAASi, and other CKD/CVD/T2D-related treatments prescribed as part of routine care will be collected. In all cases, the decision to treat a patient with dapagliflozin will be made prior to the decision to enroll a patient into the study. All treatment decisions are at the discretion of the current patient's physician, based on clinical judgment and recommendations included in the approved label and national treatment protocols, and are not mandated by this protocol.

Study measures:

* Baseline demographic, clinical characteristics, comorbidities and medications
* Post-index medications (changes, including addition, and discontinuation, and time to discontinuation for dapagliflozin)
* Post-index cardio-renal events
* Post-index healthcare resource use Sample Size Estimations: This study does not involve hypothesis testing. No formal sample size and power calculations have been performed. Across participating CEE countries (Bulgaria, Croatia, Hungary, Poland, Romania, Serbia and Slovenia), an estimated number of 1090 patients is planned for inclusion, with country target numbers varying between 70 and 300 patients, depending on preliminary feasibility with sites, the size of the country and reimbursement status at study start and during the study. The target number of patients is planned to be enrolled in 6-8 months across the region. If this target sample is not reached, this does not imply study failure, but the precision on estimates will change.

Statistical Analysis: The statistical analyses will be fully described in the Statistical Analysis Plan (SAP) as appropriate. Descriptive analyses will be performed to describe the characteristics of the cohort studied. Continuous variables will be summarized using means with standard deviations (SDs), medians with interquartile ranges (IQR), and minimum and maximum values. The number and percentages of patients will be used to summarize categorical variables, including a separate category for patients with missing data at baseline. Missing data will be quantified for all study variables, but there will be no attempts to impute them. For the secondary objective, the time to discontinuation will be estimated using the Kaplan-Meier method. Summary statistics will be used to describe proportions of patients with the event changes within the set time windows.

Baseline demographic and clinical characteristics will be summarized on the index date. For laboratory data, the value closest to index (in the last year before or on the index date) will be used. Comorbidities and medical history will be summarized in the last year before index date. Stratified analyses based on baseline demographic and clinical characteristics may be performed.

Summary statistics will be used to describe treatment patterns and drug utilisation. Further specification on planned analyses will be provided in the SAP

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥18 years) at the time of dapagliflozin start
2. Patient receives treatment with dapagliflozin for CKD in accordance with the dapagliflozin product label and local dapagliflozin reimbursement criteria for CKD

   Note: CKD diagnosis is based on the following KDIGO criteria [KDIGO 2012] that defines CKD as abnormalities of kidney structure or function, present for >3 months, with implications for health and at least one of the following criteria:
   * AER ≥30 mg/24 hours;
   * ACR ≥30 mg/g (≥3 mg/mmol);
   * eGFR <60 ml/min/1.73 m2.
3. Signed and dated informed consent prior to enrollment in the study.

Exclusion Criteria:

1. Diagnosed with type 1 diabetes [ICD-10 codes E10 and O24.0] at any time before index date.
2. Diagnosed with gestational diabetes mellitus [ICD-10 code O24.419] at any time before index date.
3. Patient is enrolled less than 30 days or more than 90 days, following initiation of dapagliflozin.
4. Prior treatment (at any time before index date) with dapagliflozin or other SGLT-2i
5. Enrolment in a clinical trial that includes specific treatments as investigational medicinal product on or 3 months before index date
6. Renal transplant at any time before index date
7. End stage renal disease (eGFR <15 ml/min/1.73m2) on index date
8. Chronic dialysis on or at any time before index date

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients with CKD who meet the country-specific label for dapagliflozin as treatment for CKD across CEE. Patients newly initiated on treatment with dapagliflozin for CKD will be eligible for enrolment by physicians from both outpatient and inpatient settings.
Sampling Method: Probability Sample
Enrollment: 1086 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Dapagliflozin utilisation: to describe characteristics among patients who are treated with dapagliflozin. | 12 months prior to the index date
  Baseline selected event rates (hospitalizations: all-cause, and cardiorenal) / number of events per year.
  Baseline concomitant medications, by drug class and specific drugs of interest
ANTHROPOMETRIC CHARACTERISTICS at study index date | 12 months prior to the index date
  Weight / kg Height / cm
CLINICAL CHARACTERISTICS | 12 months prior to the index date
  Year of initial diagnosis of CKD / year eGFR / ml/min/1.73 m2 Urine albumin-to-creatinine ratio (uACR) / mg/mmol Urine protein-to-creatinine ratio (uPCR) / mg/g

SECONDARY OUTCOMES:
To describe selected outcomes of interest and treatment patterns among CKD patients treated with dapagliflozin | 12 months after Index
  Assessment of CKD progression
  Number (events number per year), proportion (%) of patients and event rates any time within 1 year after index, related to hospitalisations (events number per year) for the following events:
  Dapagliflozin treatment patterns RAASi treatment patterns Other CKD/CVD/GLD treatment patterns
CLINICAL CHARACTERISTICS | 12 MONTHS SINCE INDEX DATE
  eGFR / ml/min/1.73 m2 Urine albumin-to-creatinine ratio (uACR) / mg/mmol Urine protein-to-creatinine ratio (uPCR) / mg/g

CONTACTS AND LOCATIONS:
Locations (56):
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Research Site, Zagreb, Croatia
- Hungary (14):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gödöllő
  - Research Site, Karcag
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nagykanizsa
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Szeged
  - Research Site, Szombathely
  - Research Site, Veszprém
- Poland (17):
  - Research Site, Bialystok
  - Research Site, Bolesławiec
  - Research Site, Bydgoszcz
  - Research Site, Choszczno
  - Research Site, Czarnków
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Opole
  - Research Site, Sieradz
  - Research Site, Szczecin
  - Research Site, Środa Wielkopolska
  - Research Site, Węgrów
  - Research Site, Wroclaw
  - Research Site, Zielona Góra
  - Research Site, Żywiec
- Romania (10):
  - Research Site, Bistriţa
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Galati
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Reşiţa
  - Research Site, Satu Mare
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Research Site, Belgrade, Serbia
- Slovenia (10):
  - Research Site, Brežice
  - Research Site, Cerknica
  - Research Site, Mengeš
  - Research Site, Portorož
  - Research Site, Ptuj
  - Research Site, Radlje ob Dravi
  - Research Site, Ruše
  - Research Site, Sevnica
  - Research Site, Škofja Loka
  - Research Site, Zagorje